CLINICAL TRIAL: NCT06998004
Title: A Phase I, Randomized, Double-blind, Multi-centre, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Reactogenicity and Immunogenicity of AstriVax' Investigational Vaccine for the Prevention of Yellow Fever (AVX70120), and of AstriVax' Investigational Vaccine for the Prevention of Rabies (AVX70481), in Healthy Adults Aged 18 to 40 Years
Brief Title: A Trial to Evaluate the Safety and Immunogenicity of an Investigational Vaccine for the Prevention of Yellow Fever, and of an Investigational Vaccine for the Prevention of Rabies, in Healthy Adults
Acronym: SAFYR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstriVax Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AVX1248-101; 2024-511194-29-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Yellow Fever; Rabies
MeSH Terms: conditions — Yellow Fever; Rabies | interventions — Floors and Floorcoverings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- AVX70120 low dose level (Experimental): Participants in this arm receive AVX70120 low dose level at Day 1
  Interventions: Biological: AVX70120 low dose level
- AVX70120 middle dose level (Experimental): Participants in this arm receive AVX70120 middle dose level at Day 1
  Interventions: Biological: AVX70120 middle dose level
- AVX70120 high dose level (Experimental): Participants in this arm receive AVX70120 high dose level at Day 1
  Interventions: Biological: AVX70120 high dose level
- AVX70481 low dose level (Experimental): Participants in this arm receive AVX70481 low dose level at Day 1
  Interventions: Biological: AVX70481 low dose level
- AVX70481 middle dose level (Experimental): Participants in this arm receive AVX70481 middle dose level at Day 1
  Interventions: Biological: AVX70481 middle dose level
- AVX70481 high dose level (Experimental): Participants in this arm receive AVX70481 high dose level at Day 1
  Interventions: Biological: AVX70481 high dose level
- Placebo (Placebo Comparator): Participants in this arm receive Placebo at Day 1
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AVX70120 low dose level — Low dose level of AVX70120, AstriVax' investigational vaccine for the prevention of yellow fever
  Arms: AVX70120 low dose level
Biological: AVX70120 middle dose level — Middle dose level of AVX70120, AstriVax' investigational vaccine for the prevention of yellow fever
  Arms: AVX70120 middle dose level
Biological: AVX70120 high dose level — High dose level of AVX70120, AstriVax' investigational vaccine for the prevention of yellow fever
  Arms: AVX70120 high dose level
Biological: AVX70481 low dose level — Low dose level of AVX70481, AstriVax' investigational vaccine for the prevention of rabies
  Arms: AVX70481 low dose level
Biological: AVX70481 middle dose level — Middle dose level of AVX70481, AstriVax' investigational vaccine for the prevention of rabies
  Arms: AVX70481 middle dose level
Biological: AVX70481 high dose level — High dose level of AVX70481, AstriVax' investigational vaccine for the prevention of rabies
  Arms: AVX70481 high dose level
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this first time in humans trial is to evaluate the safety, reactogenicity and immunogenicity of AVX70120 and of AVX70481 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between, and including, 18 and 40 years of age on the day of the Screening Visit
* Healthy individual, as established by the Investigator
* Able to read and understand the informed consent form, and written informed consent obtained from the participant
* Participants who, in the opinion of the Investigator, can and will comply with the requirements of the protocol

Exclusion Criteria:

* Body Mass Index <18.0 or >32.0 kg/m2
* Use of any investigational or non-registered product other than the study intervention within 1 month preceding study vaccination, or planned use during the study period
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or non-registered product
* Administration / planned administration of any vaccine not foreseen by the study protocol within 1 month preceding study vaccination and up to Day 31
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months preceding study vaccination, or planned chronic administration at any time during the study period
* Planned administration of long-acting immune-modifying drugs at any time during the study period
* Administration of immunoglobulins and / or any blood or blood-derived products within 3 months preceding study vaccination, or planned administration during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history, family history or physical examination
* History of or current autoimmune disease
* Personal or family history of thymic pathology
* History of any neurological disorders or seizures
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the investigational vaccines
* Malignancies or lymphoproliferative disorders within previous 5 years
* Moderate or severe acute disease in the opinion of the Investigator, and / or fever at the time of study intervention
* Alcohol, prescription drug, or substance (ab)use that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Pregnant or lactating woman
* Woman of childbearing potential who is not utilising a highly effective birth control method for at least 1 month preceding study vaccination, or planning to discontinue highly effective birth control methods during the study period.
* Participants employed by the Sponsor, by the vendors working on behalf of the Sponsor, by the Investigator or the study site, or close relatives of research staff working on this study
* Medical condition or use of medication(s) that can increase the risk of bleeding or haematoma
* Any other condition or finding that the Investigator judges may interfere with study procedures or study results

Note: other protocol-defined inclusion / exclusion criteria may apply.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-06-16 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited adverse events | During a 14-day follow-up period after vaccination
Occurrence of unsolicited adverse events | From Day 1 up to 1 month after vaccination
Occurrence of hematological and biochemical laboratory abnormalities | From Day 1 up to 6 months after vaccination
Occurrence of adverse events of special interest | From Day 1 up to 1 year after vaccination
Occurrence of serious adverse events | From Day 1 up to 1 year after vaccination

SECONDARY OUTCOMES:
Humoral immune response following administration of the investigational vaccines | From Day 1 up to 1 year after vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Centre for the Evaluation of Vaccination (CEV), Antwerp
  - University Hospital Ghent - Centrum voor Vaccinologie (CEVAC), Ghent